CLINICAL TRIAL: NCT00685984
Title: Peripheral Endothelial Function and Coronary Status in Asymptomatic Type 2 Diabetic Patients: Relations With Coronary Microcirculation Assessed With Trans-thoracic Echo-doppler
Brief Title: Peripheral Endothelial Function and Coronary Status in Asymptomatic Diabetic Patients
Acronym: PEFDIA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Alfediam (Other)
Responsible Party: Sponsor
Other Study IDs: P070403
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-05

CONDITIONS: Myocardial Ischemia
Keywords: Type 2 diabetes; silent myocardial ischemia; endothelial function
MeSH Terms: conditions — Myocardial Ischemia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1
- 2
- 3

SUMMARY:
Silent myocardial ischemia is usual in type 2 diabetic patients and associated with coronary stenoses and endothelial dysfunction or both. We therefore hypothesized that peripheral endothelial dysfunction is a marker of silent myocardial ischemia. The aim of the study is, in 120 asymptomatic type 2 diabetic patients, to evaluate the relations between coronary status, assessed with myocardial scintigraphy and subsequent coronary angiography in case of abnormality, and peripheral endothelial function, according to post-occlusive hyperaemia endothelium-dependent brachial artery dilation.

DETAILED DESCRIPTION:
Coronary microcirculation, non invasively assessed with trans-thoracic echo-doppler (coronary blood flow before and after cold pressure testing), and biochemical markers of endothelial dysfunction will also be measured. Correlations between peripheral and coronary endothelial functions will be checked. The measurements will be performed and validated in two other groups

* 30 patients with overweight but free of diabetes, matched with the patients with diabetes for age, gender and body mass index
* 30 control subjects.Reproducibility of the methods will be assessed in 10 patients of the three groups of subjects.

ELIGIBILITY:
Inclusion criteria :

FOR TYPE 2 DIABETIC PATIENTS Asymptomatic:

* with normal resting ECG
* coronary primary prevention
* other cardiovascular risk factors justifying screening for silent myocardial ischemia and coronary stenoses in case of silent myocardial ischemia.

FOR PATIENTS WITH OVERWEIGHT:

* Asymptomatic with normal resting ECG
* coronary primary prevention
* Body mass index 25-40 kg/m²
* Without diabetes.

CONTROLS Asymptomatic:

* coronary primary prevention
* Body mass index 18-25 kg/m²
* Without diabetes
* Without cardiovascular risk factors including dyslipidemia, hypertension, smoking habits, No treatment

Exclusion criteria :

* pregnancy
* renal failure
* acrosyndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * type 2 diabetes
  * overweight free of diabetes
  * control
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Post-occlusive hyperaemia endothelium-dependent brachial artery dilation | immediate

SECONDARY OUTCOMES:
noninvasive coronary microcirculation assessed with transthoracic ECHODOPPLER | immediate
cardiac autonomic neuropathy | immediate
cardiac transthoracic echography | immediate
biologic markers of endothelial function | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COSSON, MD phD, Principal Investigator — Hôpital Jean Verdier
Locations (1):
- Hôpital Jean Verdier Service of Endocrinologie-Diabétologie-Nutrition, Bondy, France

REFERENCES:
- [Result] Cosson E, Pham I, Valensi P, Paries J, Attali JR, Nitenberg A. Impaired coronary endothelium-dependent vasodilation is associated with microalbuminuria in patients with type 2 diabetes and angiographically normal coronary arteries. Diabetes Care. 2006 Jan;29(1):107-12. doi: 10.2337/diacare.29.1.107. PMID 16373905
- [Derived] Pham I, Nguyen MT, Valensi P, Rousseau H, Nitenberg A, Vicaut E, Cosson E. Noninvasive study of coronary microcirculation response to a cold pressor test. Eur J Clin Invest. 2015 Feb;45(2):135-43. doi: 10.1111/eci.12389. Epub 2015 Jan 7. PMID 25490913
- [Derived] Nguyen MT, Pham I, Valensi P, Rousseau H, Vicaut E, Laguillier-Morizot C, Nitenberg A, Cosson E. Flow-mediated-paradoxical vasoconstriction is independently associated with asymptomatic myocardial ischemia and coronary artery disease in type 2 diabetic patients. Cardiovasc Diabetol. 2014 Jan 15;13:20. doi: 10.1186/1475-2840-13-20. PMID 24428877